CLINICAL TRIAL: NCT02152709
Title: A Phase 3, Randomized, Controlled, and Blinded Clinical Trial to Evaluate Safety and Immunogenicity of 10µg/0.5ml Hepatitis B Vaccine for Infants and Other Age Groups.
Brief Title: Study of Evaluating Safety and Immunogenicity of 10µg/0.5ml Hepatitis B Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Tiantan Biological Products Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JSEPI-003
Record Dates: First submitted 2014-05-19; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis B
Keywords: Safety; Immunogenicity; Vaccine; Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10µg/0.5ml hepatitis B vaccine (Experimental): 3 dose of 10µg/0.5ml hepatitis B vaccine made by recombinant deoxyribonudeic acid techniques in saccharomyces cereviside.Produced by Beijing Tiantan Biological Products Co., Ltd. Lot number: YHB2008063S1.
  Interventions: Biological: 3 dose of 10µg/0.5ml hepatitis B vaccine
- 5µg/0.5ml hepatitis B vaccine (Active Comparator): 3 dose of 5µg/0.5ml hepatitis B vaccine made by recombinant deoxyribonudeic acid techniques in saccharomyces cereviside.Produced by Beijing Tiantan Biological Products Co., Ltd. Lot number:20080603.
  Interventions: Biological: 3 dose of 5µg/0.5ml hepatitis B vaccine

INTERVENTIONS:
Biological: 3 dose of 10µg/0.5ml hepatitis B vaccine — 3 dose of 10µg/0.5ml hepatitis B vaccine made by recombinant deoxyribonudeic acid techniques in saccharomyces cereviside were administered intramuscular injection at 0, 1, 6 momth interval.
  Arms: 10µg/0.5ml hepatitis B vaccine
Biological: 3 dose of 5µg/0.5ml hepatitis B vaccine — 3 dose of 5µg/0.5ml hepatitis B vaccine made by recombinant deoxyribonudeic acid techniques in saccharomyces cereviside were administered intramuscular injection at 0, 1, 6 momth interval.
  Arms: 5µg/0.5ml hepatitis B vaccine

SUMMARY:
The main objective of this study was to evaluate the safety and immunogenicity of 10µg/0.5ml and 5µg/0.5ml hepatitis B vaccine made by recombinant deoxyribonudeic acid techniques in saccharomyces cereviside yeast for infants and other age groups.

ELIGIBILITY:
Inclusion Criteria (For Infant Group):

* Healthy full-term infant after birth, Apgar score ≥7.
* Guardian signed informed consent.
* Guardian can comply with the requirements of the clinical trial.
* Without administering immunoglobulin during the following period.
* Axillary temperature ≤37.0 ℃.

Inclusion Criteria (For Other Age Groups):

* More than 1 month old healthy people, without the history of hepatitis B infection.
* Subjects or their guardians signed informed consent.
* After questioning medical history, physical examination and being judged as healthy subject.
* Without the history of hepatitis B vaccination.
* Subjects or their guardians can comply with requirements of the clinical trail.
* Without other prevention drugs or immunoglobulin administered within two weeks before the clinical trail or during the following period.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria (For Infant Group):

* Apgar score of infant after birth <7.
* With nervous system damage after birth, or with the family history of mental illness, epilepsy or encephalopathy.
* With immune system dysfunction.
* With vitamin deficiency.
* With acute febrile diseases, or infectious diseases.
* With congenital malformations, developmental disorders or serious chronic illness.
* With thrombocytopenia or other coagulation disorders.
* Administered immunoglobulin during the period of the clinical trail, especially administered Hepatitis B immunoglobulin to the infant of Hepatitis B infected mother.
* With endemic disease.
* Participate another clinical trial during the period of the clinical trail.
* Any circumstance that may affect clinical trail evaluation.

Exclusion Criteria (For Other Age Groups):

* With allergies, seizures, epilepsy, encephalopathy or with family history of mental illness.
* Allergic to any component of the study vaccine.
* With immune system dysfunction.
* Hepatitis B infected people.
* Anti-HBs was positive screened by ELISA kit.
* Either anti-HBs ≥10mIU/ml or HBsAg was positive screened by Radioimmunoassay method.
* With acute febrile diseases or infectious diseases.
* With congenital malformations, developmental disorders or serious chronic illness.
* With thrombocytopenia or other coagulation disorders.
* With the history of severe allergic reactions.
* Administered other prevention drugs or immunoglobulin within two weeks before the clinical trail or during the following period.
* With any acute illness that requires antibiotics or anti-viral treatment within 7 days before the clinical trail.
* With vitamin deficiency.
* With the history of febrile convulsion.
* Axillary temperature ≥38.0 ℃ within 3 days before the clinical trail.
* Participate another clinical trial during the period of the clinical trail.
* Pregnant woman.
* Any circumstance that may affect clinical trail evaluation.

Ages: 1 Day to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Within 28 days after hepatitis B vaccination
  To analyze the number of subjects with adverse events within 28 days after administered each of hepatitis B vaccine.
Geometric mean concentration of anti-hepatitis B virus surface antigen antibody | The 28th day after whole course of hepatitis B vaccination
  Geometric mean concentration of anti-hepatitis B virus surface antigen antibody was measured by chemiluminescence assay and expressed with mIU/mL.

SECONDARY OUTCOMES:
The rate of hepatitis B virus perinatal transmission | The 28th day after whole course of hepatitis B vaccination
  To analyze the rate of hepatitis B virus perinatal transmission after whole course of hepatitis B vaccination.
Geometric mean concentration of anti-hepatitis B virus surface antigen antibody after the second dose of hepatitis B vaccination | The 28th day after the second of hepatitis B vaccination
  Geometric mean concentration of anti-hepatitis B virus surface antigen antibody was measured by chemiluminescence assay and expressed with mIU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Fubao Ma, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Kang G, Ma F, Chen H, Yang Y, Guo S, Wang Z, Liang X, Li L, Cui F, Zhang L. Efficacy of antigen dosage on the hepatitis B vaccine response in infants born to hepatitis B-uninfected and hepatitis B-infected mothers. Vaccine. 2015 Aug 7;33(33):4093-9. doi: 10.1016/j.vaccine.2015.06.081. Epub 2015 Jul 3. PMID 26144895